CLINICAL TRIAL: NCT01927809
Title: Genetics of Hirschsprung's Disease - Can Genetic Mosaicism Due to Early Somatic Mutations, Explain Disease Development?
Brief Title: Genetic Mosaicism in Hirschsprung's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, R. Garritsen, MD, Erasmus Medical Center
Other Study IDs: NL42585.078.12
Record Dates: First submitted 2013-07-08; First posted 2013-08-23 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Hirschsprung Disease
Keywords: Hereditary Diseases; Colon
MeSH Terms: conditions — Hirschsprung Disease; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, skin tissue, colon tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
Hirschsprung's disease is a complex genetic disorder. The etiology of this disease is not completely understood. It is characterized by the absence of ganglia (nerve cells) in de distal colon. This impairs bowel relaxation which can lead to bowel disfunction, toxic megacolon, ileus and enterocolitis. So far, several genes have been identified that play a role in Hirschsprung's disease. The precise mechanisms however, remain unclear. This study wants to identify new mutations and hopefully clarify more about the etiology of the disease.

ELIGIBILITY:
Inclusion Criteria:

* All children with Hirschsprung's disease that will receive a corrective pull through procedure

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients will be selected in the two participating hospitals. The Erasmus MC - Sophia Children's hospital and the UMC St. Radboud.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-04; Primary Completion 2020-12 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
New somatic mutation | During surgery (coolection); after inclusion of approx. 25 patients (preliminairy analysis); final analysis after end of the study (approx. 3 years from first inclusion)
  Primary outcome measure of this study is to identify new (previously unknown) somatic mutations as a cause for the development of Hirschsprung's disease. Tissue to find these mutations will be gathered during surgery for all patients (see protocol). When sufficient samples are collected (est 25 samples) a first comparative analysis for new somatic mutations will be performed. After the end of the study a final analysis for new somatic mutation will be performed.

SECONDARY OUTCOMES:
Correlation disease type | At the end of the study (approximately 3 years after inclusion of first patient)
  Secondary outcome measure is to assess if any of the found mutations can be correlated with the type of Hirschsprung's disease (i.e. long-segment, short segment). This will be done after all patients DNA is analysed for somatic mutations after closure of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Rhiana Garritsen, MD, Principal Investigator — Erasmus MC - Sophia; Katherine MacKenzie, Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - UMC St Radboud, Nijmegen, Gelderland
  - Erasmus Medical Center - Sophia, Rotterdam, South Holland